CLINICAL TRIAL: NCT07391176
Title: Evaluation of the Effectiveness of Deep Intervention in the Submental Region in Context of Managing of Double Chin (Clinical Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tishreen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tishreen-U O,M Fascial surgery
Record Dates: First submitted 2026-01-20; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Evaluation of Deep Plan Intervention in the Submental Region for Double Chin Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical submental correction for Double chin (Experimental)
  Interventions: Procedure: Evaluation of platysma muscle partial resection with midline plication for double chin correction

INTERVENTIONS:
Procedure: Evaluation of platysma muscle partial resection with midline plication for double chin correction — The surgical procedure will be performed in two consecutive stages
  Phase one - midline correction:
  1. submental liposuction : fat is aspirated from the submental region via a small puncture using a cannula.
  2. Access expansion: the puncture entry is extended to form a small horizontal submental incision.
  3. Dissection and exposure: the area is dissected through this incision using blunt dissection techniques to expose the midline platysma muscle.
  4. Muscle excision: an elliptical segment of the platysma muscle is excised at the midline level.
  5. Closure: the resulting muscular defect is closed with primary suturing.
  Phase two-lateral correction :
  1. lateral access :the lateral aspect of the platysma muscle and the superficial musculoaponeurotic system is accessed via concealed peri-auricular incision
  2. Plication and tightening: the platysma and smas are plicate and tighten along natural tension lines to lift the jawline and neck contours.
  3. finally redundant skin excision and suturing.

SUMMARY:
what problem is this study investigating some people suffer from what is called a double chin or the accumulation of fat and sagging skin under the chin which may affect the profile and cause dissatisfaction what is the main objective of this study this study aims to evaluating the efficacy and safety of a targeted submentoplasty surgical procedure. this procedure involves

* making a horizontal submental incision
* performing midline platysma resection and suturing with lateral platysma plication along defined vectors
* Excision of redundant skin potentially extending to the periauricular area as needed.

Who can participate in this study inclusion criteria

* Be 45 years of age or older
* present with moderate to severe submental fullness and skin laxity classified as Dedo type D(prominent platysma bands with significant skin redundancy)
* Be in good general systemic health with no contraindication to elective surgery or anesthesia.
* Have a stable weight (no significant gain or loss in the past 6 months). .Express dissatisfaction with their submental contour and desire surgical correction.
* Be anon-smoker or agree to cease smoking for a minimum of 4 weeks before and after the procedure.

Exclusion criteria

* previous history of any surgical procedure in the submental area,neck,or lower face(face lift ,neck lift, submentoplasty ,or liposuction).
* previous history of any injectable treatment (deoxycholic acid ,filler, collagen stimulators ) in the submental area within the past 12 months.
* presence of an active skin infection or inflammatory condition in the treatment area.
* Known bleeding disorder or use of anticoagulant medication that cannot be safely paused for the procedure.
* unrealistic expectations regarding surgical outcomes.
* Significant medical comorbidities that increase surgical risk(uncontrolled diabetes ,severe cardiovascular disease).

Final eligibility will be determined during a comprehensive screening consultation with the principal surgeon, which will include a physical examination and detailed medical history review.

What does the study involved if you participate? This is a prospective ,singal-arm clinical study designed to evaluate the effectiveness and safety of a targeted submentoplasty procedure. A total of 12 eligible female participants will be enrolled.

procedure details : if you qualify and consent to participate ,you will undergo the following surgical intervention:

* The procedure will be performed under local anesthesia or general anesthesia.
* It involves : making a horizontal submental incision ,performing midline platysma resection and suturing , lateral platysma plication along defined vectors , and excision of redundant skin with possible periauricular extension.
* The surgery will be performed in latakia university hospital.

Study time line and Assessments:

Your participation will involve the following schedule:

* Pre-Treatment visit: A screening visit to confirm eligibility , take detailed medical history , and perform standardized photographic documentation(front and side views) of your face and neck.
* The treatment visit :The day of the scheduled surgical procedure.
* Follow-up visit : You will be required to attend post-operative follow-up appointments at two key time points to monitor results and safety :
* 1 month after the procedure.
* 3 month after the procedure.

Assessments at Each follow-up: Each follow-up visit will include:

* Photographic documentation : Repeated standardized photographs (identical views to the pre-treatment photos) to allow for objective comparison and assessment of improvement .
* Clinical Evaluation : An assessment by the surgeon for healing , aesthetic outcome , and any potential complication .
* Patient-repoted outcomes :you will be asked to complete a brief questionnaire about your satisfaction with the results , improvement in your appearance , and any symptoms .
* Your commitment:

participation requires your commitment to attend the pre-treatment visit , undergo the surgery , and attend both follow-up visits at 1 month 3 months post-operative care instructions provided by the surgical team.

. Data collection: The primary method for evaluating effectiveness will be the comparative analysis of the standardized photographs taken before the surgery and at the 1-month and 3-moths follow-up visits. clinical notes and your questionnaire responses will provide supporting data on safety and satisfaction.

. What are the expected benefits of participation? you may achieve an improved appearance and definition of the chin area through surgical procedure. this can enhance facial harmony and potentially boost your self-confidence.

What are the potential risks of participation? potential risks associated with this surgical procedure include, but are not limited to: bleeding, infection, noticeable scarring, adverse reactions to anesthesia, temporary or permanent nerve damage, irregularity in the jawline and neck contour changes in ear position

ELIGIBILITY:
Inclusion Criteria:

1. Age: 45 years and older.
2. Systemic health : systemically healthy individuals (without significant systemic diseases), in good general health (ASA SCORE I OR II).
3. Anatomical classification: participants classified as Type D according to Dedo Cervicomental angle classification (characterized by increased submental fat with platysma laxity and loss of angle definition due to both skin and fat).
4. weight stability : proposed addition. stable weight loss.

Exclusion Criteria:

1. Age: under 45 years
2. Systemic diseases: presence of uncontrolled or relevant systemic diseases affecting wound healing or outcomes

   * active autoimmune diseases
   * uncontrolled diabetes mellitus.
   * bleeding or coagulation disorders
   * advanced chronic liver or kidney disease.
3. anatomical classification: any Dedo classification other than type D (Type A,B,C).
4. Relevant medical history :proposed addition.

   * history of previous surgical or cosmetic interventions in the neck/chin area
   * active skin diseases or infections in the treatment area. .known history of hypertrophic or keloid scarring.
5. Medication and supplements: proposed addition.

   * use of anticoagulant medications (warfarin, clopidogrel)
   * use supplements or medications affecting bleeding (high-dose aspirin, ibuprofen, fish oil, garlic ,ginkgo biloba) within a specified period before the procedure.
6. Lifestyle factors: proposed addition.

   * heavy smoking ( negatively affects wound healing ).
   * significant alcohol consumption.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-01-09 (Actual); Primary Completion 2026-01-10 (Actual); Study Completion 2026-01-19 (Actual)

PRIMARY OUTCOMES:
Cervicomental angle (in degrees) as measured using AutoCAD software. | Measured at three time point : before treatment(baseline),1 month after treatment, and 3 moths after treatment.
  The chin point( the lowest point on the chin in lateral view) and a point on the sternum(the highest prominent point of the sternum at the head) will be identified.
  Then, the point of the chin-neck junction(the lowest point of the curvature under the chin) will be determined. Subsequently, a line will be drawn connecting the chin point to the chin-neck junction point (the first side),and another line connecting the chin-neck junction point to sternum point(the second side) using the line tool in Adobe Photoshop. finally, the angel formed between these two sides will be measured using AutoCAD program.

CONTACTS AND LOCATIONS:
Locations (1):
- Latakia university, Latakia, Syria

IPD SHARING:
Plan to Share IPD: No